CLINICAL TRIAL: NCT07331532
Title: PET Imaging Study of 68Ga-PFA2 Probe for Annexin A2-Positive Tumors
Brief Title: 68Ga-PFA2 PET Imaging for the Diagnosis of Annexin A2-Positive Tumors
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Tingting Yuan, Attending physician, Peking University First Hospital
Other Study IDs: PFA2 001
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms、Lung Neoplasms、Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patients will undergo PET/CT imaging with 68Ga-PFA2 to assess metastasis detection.

SUMMARY:
Tumor metastasis and invasion are the leading causes of cancer-related deaths, with over 90% of cancer patients dying from distant metastasis. Tumor cells spread to distant organs through local infiltration, hematogenous metastasis, or lymph node metastasis, complicating treatment and severely affecting the prognosis and survival rate of patients. Therefore, precise and early assessment of tumor invasion and metastasis is crucial for optimizing personalized treatment plans and improving patient survival.

Currently, the detection of tumor metastasis primarily relies on imaging examinations, blood biomarkers, and histopathological analysis. Among these, 18F-FDG PET/CT plays a key role in tumor staging and distant metastasis evaluation. However, its sensitivity is low for certain tumors, such as well-differentiated hepatocellular carcinoma, colorectal cancer, and glioblastoma, and factors like inflammation can lead to false positives. Additionally, serum tumor markers (such as AFP, CEA, and CA19-9) often lack specificity in some patients, and histopathological analysis requires invasive sampling, making real-time monitoring difficult. Therefore, the development of non-invasive methods based on molecular targets for early and precise detection of tumor invasion and metastasis holds significant clinical value.

Tumor invasion and metastasis is a complex process involving multiple molecules that drive cancer cell proliferation, invasion of surrounding tissues, and the formation of secondary tumors in distant organs. During invasion and metastasis, cancer cells are often subjected to mechanical stress, such as compression and shear forces, making the repair of cell membrane damage crucial for the survival of invasive cancer cells. Annexin A2 (ANXA2) is a multifunctional protein that plays a key role in cancer cell membrane repair, proliferation, migration, invasion, and metastasis. Studies have shown that silencing ANXA2 or inhibiting its function with neutralizing antibodies reduces the ability of cancer cells to repair membrane damage, thereby limiting tumor cell dissemination. Abnormal expression of ANXA2 is a common feature in many types of tumors. The expression level of ANXA2 in tumors is closely associated with the growth, invasion, and metastasis of pancreatic cancer, colorectal cancer, breast cancer, gliomas, and other tumors.

Furthermore, ANXA2 promotes tumor cell proliferation by facilitating DNA replication, cell cycle progression, and neovascularization, thereby supporting tumor growth and progression. For instance, in breast cancer, ANXA2 promotes STAT3 activation through Tyr23 phosphorylation, upregulating cyclin D1 and MMP2/9, which accelerates breast cancer proliferation, invasion, and metastasis. In pancreatic cancer, ANXA2 regulates the Src/ANXA2/STAT3 signaling pathway to promote epithelial-mesenchymal transition (EMT), enhancing cellular invasiveness. In non-small cell lung cancer (NSCLC), ANXA2 overexpression correlates with tumor staging, lymph node metastasis, and distant metastasis, and can serve as an independent prognostic marker. In hepatocellular carcinoma (HCC), high ANXA2 expression is not only associated with higher tumor recurrence rates but also promotes angiogenesis, further driving tumor progression. In glioblastoma (GBM) and colorectal cancer, ANXA2 has also been shown to accelerate disease progression through mechanisms such as extracellular matrix degradation, angiogenesis, and tumor microenvironment regulation.

ANXA2 not only serves as a poor prognostic factor for various cancers but also holds potential as a therapeutic target. Several monoclonal antibodies targeting ANXA2 have shown significant antitumor and antiangiogenic effects. Rajkumar et al. demonstrated that the monoclonal antibody mAb150, targeting the N-terminal epitope of ANXA2, enhances cancer stem cells' re-entry into the cell cycle, reducing migration and EMT in activated cancer cells, ultimately inhibiting ascites formation and extending survival in a mouse ovarian cancer model. Another monoclonal antibody, ch2448, targets the unique glycan epitope of ANXA2, triggering antibody-dependent cell-mediated cytotoxicity, effectively inhibiting tumor formation and delaying or preventing teratoma development. In addition to large molecular antibodies, the first small-molecule inhibitor of ANXA2 in triple-negative breast cancer, 5α-epoxyalantolactone (5-EAL), has been discovered. 5-EAL selectively binds to the conserved cysteine residue of ANXA2, inhibiting the formation of the ANXA2-S100A10 heterotetramer complex, effectively suppressing TNBC proliferation and metastasis. These findings highlight the enormous diagnostic and therapeutic potential of ANXA2 as a biomarker for malignant cancers.

Given the high expression of ANXA2 in various tumors and

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years.
* Diagnosed with confirmed lung cancer.
* Scheduled to undergo pathological tissue biopsy or surgical treatment within the next two months.
* Able to fully comprehend and voluntarily participate in the study.
* Able to provide informed consent.
* Capable of cooperating independently to complete the examinations.

Exclusion Criteria:

* Patients with other malignancies or severe comorbidities that affect their ability to participate.
* Patients unable to provide informed consent due to cognitive impairment.
* Patients with contraindications to PET/CT scans or 68Ga-PFA2 administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include lung cancer patients, both suspected and confirmed, who are scheduled to undergo PET/CT imaging using the 68Ga-PFA2 probe. The study will focus on patients aged 18-80 years with confirmed lung cancer, and the participants should be able to understand the study protocol, provide informed consent, and cooperate with examination procedures.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of 68Ga-PFA2 PET Imaging in Detecting Metastasis in Lung Cancer | Primary data collection will be completed at the end of the study, with imaging performed at baseline and 30-minute, 60-minute intervals post-injection.
Diagnostic Performance of 68Ga-PFA2 PET Imaging in Detecting Metastasis in Lung Cancer | Primary data collection will be completed at the end of the study, with imaging performed at baseline and 30-minute, 60-minute intervals post-injection.
  This outcome measure evaluates the ability of the 68Ga-PFA2 PET imaging probe to detect metastases in lung cancer patients, focusing on Annexin A2-positive tumors. The primary objective is to assess its diagnostic performance compared to the standard 18F-FDG PET/CT imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university first hospital nuclear medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang Y, Jia M, Yang X, Han H, Hou G, Bi L, Yang Y, Zhang R, Zhao X, Peng C, Ouyang X. Annexin A2: The diversity of pathological effects in tumorigenesis and immune response. Int J Cancer. 2022 Aug 15;151(4):497-509. doi: 10.1002/ijc.34048. Epub 2022 May 6. PMID 35474212
- [Result] Wang YQ, Zhang F, Tian R, Ji W, Zhou Y, Sun XM, Liu Y, Wang ZY, Niu RF. Tyrosine 23 Phosphorylation of Annexin A2 Promotes Proliferation, Invasion, and Stat3 Phosphorylation in the Nucleus of Human Breast Cancer SK-BR-3 Cells. Cancer Biol Med. 2012 Dec;9(4):248-53. doi: 10.7497/j.issn.2095-3941.2012.04.005. PMID 23691485
- [Result] Foley K, Rucki AA, Xiao Q, Zhou D, Leubner A, Mo G, Kleponis J, Wu AA, Sharma R, Jiang Q, Anders RA, Iacobuzio-Donahue CA, Hajjar KA, Maitra A, Jaffee EM, Zheng L. Semaphorin 3D autocrine signaling mediates the metastatic role of annexin A2 in pancreatic cancer. Sci Signal. 2015 Aug 4;8(388):ra77. doi: 10.1126/scisignal.aaa5823. PMID 26243191
- [Result] Wirtz D, Konstantopoulos K, Searson PC. The physics of cancer: the role of physical interactions and mechanical forces in metastasis. Nat Rev Cancer. 2011 Jun 24;11(7):512-22. doi: 10.1038/nrc3080. PMID 21701513
- [Result] Cleary AS, Leonard TL, Gestl SA, Gunther EJ. Tumour cell heterogeneity maintained by cooperating subclones in Wnt-driven mammary cancers. Nature. 2014 Apr 3;508(7494):113-7. doi: 10.1038/nature13187. PMID 24695311
- [Result] Chen L, Qin G, Liu Y, Li M, Li Y, Guo LZ, Du L, Zheng W, Wu PC, Chuang YH, Wang X, Wang TD, Ho JA, Liu TM. Label-free optical metabolic imaging of adipose tissues for prediabetes diagnosis. Theranostics. 2023 Jun 19;13(11):3550-3567. doi: 10.7150/thno.82697. eCollection 2023. PMID 37441598
- [Result] Ma L, Yu H, Zhu Y, Xu K, Zhao A, Ding L, Gao H, Zhang M. Isolation and proteomic profiling of urinary exosomes from patients with colorectal cancer. Proteome Sci. 2023 Feb 9;21(1):3. doi: 10.1186/s12953-023-00203-y. PMID 36759883
- [Result] Orsaria P, Chiaravalloti A, Fiorentini A, Pistolese C, Vanni G, Granai AV, Varvaras D, Danieli R, Schillaci O, Petrella G, Buonomo OC. PET Probe-Guided Surgery in Patients with Breast Cancer: Proposal for a Methodological Approach. In Vivo. 2017 Jan 2;31(1):101-110. doi: 10.21873/invivo.11031. PMID 28064227
- [Result] Ganesh K, Massague J. Targeting metastatic cancer. Nat Med. 2021 Jan;27(1):34-44. doi: 10.1038/s41591-020-01195-4. Epub 2021 Jan 13. PMID 33442008